CLINICAL TRIAL: NCT01377974
Title: Randomized Clinical Trial of Miltefosine to Treat Mucosal Leishmaniasis at Federal District, Brazil
Brief Title: Clinical Trial of Miltefosine to Treat Mucosal Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Juliana Silva, Dr. Juliana Silva, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MILTHUB
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Leishmaniasis; Leishmaniasis, Mucocutaneous
Keywords: Leishmaniasis; Mucocutaneous Leishmaniasis; Therapeutics; meglumine antimoniate; miltefosine
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Mucocutaneous | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (Active Comparator): Meglumine antimoniate as recommended by the Brazilian Ministry of Health
  Interventions: Drug: Standard Treatment Meglumine antimoniate
- Tested Intervention (Experimental): Miltefosine as the tested intervention
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — 1 Capsule of 50mg, taken orally 2 times a day for 28 days
  Other Names: Impavido
  Arms: Tested Intervention
Drug: Standard Treatment Meglumine antimoniate — 20mgKg daily intravenous Meglumine antimoniate as oriented by the Brazilian Ministry of Health
  Other Names: pentavalent antimonial
  Arms: Standard Treatment

SUMMARY:
The purpose of this study is to determine whether miltefosine is effective in the treatment of mucosal leishmaniasis compared to meglumine antimoniate, the standard treatment.

DETAILED DESCRIPTION:
Mucosal leishmaniasis is a rare form of the disease, that affects only 6% of the patients with cutaneous leishmaniasis in the New World. It causes deformities and may be lethal if not treated. It is part of the neglected tropical diseases because on the past sixty years there was few progress regarding other treatment options or improvement at quality of life of its patients. Also, there was little interest from the pharmaceutical industry and government authorities to develop new researches. The standard treatment, meglumine antimoniate, is toxic, invasive, requires trained personnel and has many adverse effects and restrictions. On the other hand, miltefosine is the first oral drug to demonstrate efficacy against mucocutaneous leishmaniasis. Few clinical trials have being performed in Central and South American countries, but so far, just one involved mucosal leishmaniasis patients, and compared miltefosine to amphotericin B. None studies comparing its efficacy to the standard treatment have being done.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mucosal leishmaniasis
* Not previously treated, or last treatment must have occurred more than 6 months before the enrollment on the study
* Use of contraceptive method, if female on child bearing age
* Sign the agreement and consent form

Exclusion Criteria:

* Previous leishmanicidal treatment on the past 6 months before the enrollment on the study
* Electrocardiogram abnormalities on the pretreatment exams
* Previous kidney, liver and/or heart diseases
* Diabetes Mellitus
* Hypersensitivity to miltefosine or meglumine antimoniate
* Pregnant women or breastfeeding mothers
* Hiv patients

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cure | 6 months
  Re-epithelizations of mucosal ulcers or regression of symptoms

SECONDARY OUTCOMES:
Adverse effects | 6 months
  laboratory tests of blood, kidney, liver and cardiac functions, partients will be asked about nausea, vomiting, diarrhea, myalgia, or other symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Juliana SF Silva, MD, Principal Investigator — University of Brasilia; Raimunda NR Sampaio, PhD, Study Chair — University of Brasilia
Locations (1):
- Brasilia University Hospital, Brasília, Federal District, Brazil